CLINICAL TRIAL: NCT02217761
Title: Pharmacokinetic Study in Patients Receiving Posaconazole Therapy in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201112163RID
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Pharmacokinetics; Posaconazole
Keywords: Pharmacokinetics; Antifungal Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum. white cells, saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the factors influencing pharmacokinetic and pharmacodynamic properties of new antifungal agent, posaconazole in Taiwanese patients.

DETAILED DESCRIPTION:
Invasive fungal infection (IFI) may cause high mortality and morbidity in immune- compromised patients. Posaconazole, a new triazole antifungal agent with broad spectrum coverage, was approved for both treatment and prophylaxis of IFIs. Previous studies have demonstrated the relationship between posaconazole plasma concentration and efficacy, thus, the importance of posaconazole therapeutic drug monitoring (TDM) was gradually accepted. However, studies found inter- and intra-individual variation between concentrations, and these phenomenons were affected greatly by GI function, food intake and concomitant medication. Furthermore, there's a lack of posaconazole TDM study in Asian population.

The study was designed to describe the prescribing pattern of posaconazole, to study the relationship between concentration and clinical outcomes/ adverse events, to identify factors that influence plasma concentration, and to evaluate whether routine TDM is needed in our institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving posaconazole therapy
* Patients aged 13 years old or more

Exclusion Criteria:

* No posaconazole plasma concentration available

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in National Taiwan University receiving posaconazole
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-03; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Plasma posaconazole concentration | 7-10 days after taking posaconazole

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Wen Lin, Pharm. D., Principal Investigator — Graduate institute of clinical pharmacy at National Taiwan University